CLINICAL TRIAL: NCT03170414
Title: A Prospective Observational Study of Solid Organ Transplantation Utilizing HIV-Positive Donors in HIV-Positive Recipients
Brief Title: Observational Study of Solid Organ Transplantation Utilizing HIV-Positive Donors in HIV-Positive Recipients
Status: Completed | Type: Observational
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Other Study IDs: SURG-2017-24985
Record Dates: First submitted 2017-05-23; First posted 2017-05-31 (Actual); Last update posted 2024-02-12 (Actual); Status verified 2024-02

CONDITIONS: HIV; Awaiting Organ Transplant
Keywords: HIV; Kidney Transplant; Liver Transplant; Transplant; HOPE Act

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- HIV D+/R+: HIV+ recipients who receive an organ transplant from an HIV+ donor

SUMMARY:
The primary objective of this study is to evaluate the safety of solid organ transplantation using HIV-positive deceased donors (liver, kidney) and HIV-positive living donors (liver) in HIV-positive recipients.

HIV-positive individuals who agree to accept and receive a solid organ transplant from and HIV-positive donor will be followed to determine the safety and efficacy of this practice.

DETAILED DESCRIPTION:
This is a prospective observational study of solid organ transplantation utilizing HIV-positive donors in HIV-positive recipients. Stable HIV-infected adults in need of a solid organ transplant (kidney, liver) who meet standard and study specified HIV criteria for organ transplantation will be offered enrollment in the study. Deceased donors (kidney, liver) and living donors (liver) will be utilized in this protocol. No living kidney donors will be enrolled.

This study will evaluate overall survival and graft survival. In addition the study will assess potential complications of organ transplant using HIV+ donor organs, including but not limited to: HIV disease progression, development of antiretroviral resistance mutations, incidence of opportunistic infections, incidence of transplant complications, impacts of liver regeneration, incidence of viral-related malignancies, and incidence of HIV-superinfection.

ELIGIBILITY:
RECIPIENT ELIGIBILITY CRITERIA HIV-Positive Recipient Inclusion Criteria (liver, kidney)

1. Participant is able to understand and provide informed consent.
2. Participant meets standard listing criteria for transplant.
3. Documented HIV infection (by any licensed ELISA and confirmation by Western Blot, positive HIV ab IFA, or documented history of detectable HIV-1 RNA).
4. Participant is ≥ 18 years old.
5. No evidence of active opportunistic complications of HIV infection.
6. Participant CD4+ T-cell count is >/= 200/µL within 16 weeks prior to transplant for kidney transplant recipients. For liver transplant recipient, CD4+ T-cell counts need to be >/= 100/ul (or >/= 200/µL if history of opportunistic infection) within 16 weeks prior to transplant.
7. Participant most recent HIV-1 RNA < 50 copies/mL (by any FDA-approved assay performed in CLIA-approved laboratory), in the 26 weeks prior to transplant. Participants unable to tolerate ART due to organ failure or who have only recently started ART may have detectable viral load and still be considered eligible if the study team is confident there will be a safe, tolerable, and effective antiretroviral regimen once organ function is restored after transplantation.
8. Concurrence by the study team that based on medical history and ART, viral suppression can be achieved in the recipient post-transplant.
9. No history of primary CNS lymphoma or progressive PML.
10. On a stable antiretroviral regimen. Participants unable to tolerate ART due to organ failure may still be considered eligible if the study team is confident there will be a safe, tolerable, and effective antiretroviral regimen once organ function is restored after transplantation.

HIV-Positive Recipient Exclusion Criteria (liver, kidney)

1. Participant has concomitant conditions that, in the judgment of the investigators, would preclude transplantation or immunosuppression.

DONOR ELIGIBILITY CRITERIA HIV-Positive Deceased Donor (liver, kidney)

1. Must meet all clinical criteria for HIV-uninfected organ donors.
2. No evidence of invasive opportunistic complications of HIV infection.
3. Pre-implant donor organ biopsy showing no disease process that would put the recipient at increased risk of rapid progression to end-stage organ failure, to be stored for the duration of the study.
4. Donor has documented HIV infection (by any licensed ELISA and confirmation by Western Blot, positive HIV ab IFA, or history of detectable HIV-1 RNA) from a CLIA-approved laboratory.
5. If known history of HIV infection and prior antiretroviral therapy, the study team must describe the anticipated post-transplant antiretroviral regimen to be prescribed for the recipient and justify its conclusion that the regimen will be safe, tolerable and effective.

HIV-Positive Living Donor (liver)

1. Donor meets all clinical criteria to be a living liver donor other than being HIV positive.
2. Donor has documented HIV infection (by any licensed ELISA and confirmation by Western Blot, positive HIV ab IFA, or history of detectable HIV-1 RNA) from a CLIA-approved laboratory.
3. No evidence of invasive opportunistic complications of HIV infection
4. Donor CD4+ T-cell count is >/= 500/µL in the 26 weeks prior to donation.
5. The most recent HIV-1 RNA has been below 50 copies RNA/ml in the 26 weeks prior to donation.
6. On a stable antiretroviral regimen.
7. Must be evaluated by the HIV/Transplant Infectious Diseases team to verify resistance history and current ART regimens. The potential for transmission of resistant strain of HIV will be assessed.
8. Pre-implant donor liver biopsy to be stored for the duration of the study showing no evidence of a disease process that would put the donor at increased risk of progressing to end-stage organ failure after donation, or that would present a risk of poor graft function to the recipient.
9. Must be evaluated by an independent HIV study living donor advocate separate from the transplant service in addition to the living donor advocate seen by all living donors.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Stable HIV-infected adults in need of a solid organ transplant (kidney, liver) who meet standard and study specified HIV criteria for organ transplantation will be offered enrollment in the study. Deceased donors (kidney, liver) and living donors (liver) will be utilized in this protocol. No living kidney donors will be enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2017-06-15 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2023-12-01 (Actual)

PRIMARY OUTCOMES:
Patient Survival | One Year
  Patient survival at one year.

SECONDARY OUTCOMES:
Graft Survival | Months 3, 6, 9, Years 1, 2, 3
Incidence and Severity of Graft Rejection | Through study completion, up to three years
HIV Disease Progression | Through study completion, up to three years
Development of antiretroviral resistance mutations and/or X4 tropic virus in blood and allograft | Through study completion, up to three years
Incidence of bacterial, fungal, viral and other opportunistic infections | Through study completion, up to three years
Incidence of other transplant complications (surgical and vascular) | Through study completion, up to three years
Liver transplant recipients: Impact on liver regeneration | Through study completion, up to three years
Analysis of recurrent HIV associated nephropathy among kidney transplant recipients | Through study completion, up to three years
Incidence of other viral-related malignancies (HPV, EBV, HBV, HCV) | Through study completion, up to three years
Incidence of systemic HIV-superinfection in blood | Through study completion, up to three years
Incidence of tissue specific HIV-superinfection | Through study completion, up to three years

CONTACTS AND LOCATIONS:
Overall Officials: Timothy Pruett, MD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota Medical Center, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: Undecided